CLINICAL TRIAL: NCT05733052
Title: Pubourethral Plication Procedure (PPP) Cures Stress Urinary Incontinence Without Tapes- First Report.
Brief Title: Pubourethral Ligament Plication for the Surgical Treatment of Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, AHMET AKIN SIVASLIOĞLU, Professor, Muğla Sıtkı Koçman University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11/VII
Record Dates: First submitted 2022-12-27; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Urinary Incontinence; Pelvic Floor Disorders
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polyester suture arm (Experimental): A No 3 polyester suture will be inserted into the external urethral ligament, into the uurethral part of pubourethral ligament and into the pubic part of the pubourethral lgament then will be tied, but not tightly. The interventions will be carried on either side of the urethra that will be opened up by an 2.5 cm incision in the periurethral sulci.
  Interventions: Other: Polyester suture

INTERVENTIONS:
Other: Polyester suture — A No2 polyester suture will be used for tying special anatomical structures fr telieving the symptom. of stress urinary incontinence

SUMMARY:
To test efficacy and safety at six months of the proposed Pubourethral Plication Procedure (PPP) for cure of stress urinary incontinence - reinforcing pubourethral ligaments (PUL) with large diameter polyester sutures.

DETAILED DESCRIPTION:
Full thickness vaginal incisions will be made in the suburethral sulci extending from bladder neck to urethral meatus. The operation space is 2.5cm2 space. A No2 or 3 polyester suture will be inserted into PUL, immediately lateral to midurethra, into PUL origin, external urethral ligament, laterally into m.pubococcygeus, then will be tied, but not tightly. The vaginal incisions will be closed with vicryl sutures. All women will be discharged on day of surgery. During the regular follow ups the healing at stress urinary incontinence will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Urine loss on coughing controlled by hemostat behind symphysis

Exclusion Criteria:

* No exclusion criteria

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 36 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Curing effect of the suturation | 6 months
  The plication of pubourethral ligaments with a polyester suture will lead to a neoligament formation; so that the pubourethral ligaments will get strenghened. If the pubourethral ligaments get strengthened woman will not loose urine upon stressful activities such as coughing. Hence the stress test will be negative. And the rate of negative stress test within the cohort will show us the efficinecy of operation in curing urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: AHMET AKIN SIVASLIOGLU, Prof, Principal Investigator — Mugla SITKI KOÇMAN UNİVERSITY
Locations (1):
- Muğla Training and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No